CLINICAL TRIAL: NCT07356778
Title: An Open-label, Randomized, Controlled Trial to Evaluate the Efficacy of Sotatercept Add-on Therapy Compared to Standard PAH Therapy With Pulmonary Vasodilators for Pulmonary Arterial Hypertension Associated With Pulmonary Vasodilator-resistant, Unrepaired Congenital Shunts (ASD, VSD, PDA) Including Eisenmenger Syndrome：SuMILE Trial
Brief Title: A Study of Sotatercept for Patients With Eisenmenger Syndrome or Unrepaired Shunt-Associated Pulmonary Arterial Hypertension Resistant to Vasodilator Therapy
Acronym: SuMILE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kazuya Hosokawa (Other)
Responsible Party: Sponsor-Investigator, Kazuya Hosokawa, Associate professor, Center for Advanced Medical Innovation, Kyushu University, Kyushu University
Organization: Kyushu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTR-2025-Sep
Record Dates: First submitted 2025-09-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Eisenmenger Syndrome; Pulmonary Arterial Hypertension of Congenital Heart Disease
Keywords: Eisenmenger syndrome; pulmonary arterial hypertension; Congential heart disease; sotatercept
MeSH Terms: conditions — Eisenmenger Complex; Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sotatercept add-on + vasodilator-based PAH therapy (Experimental)
  Interventions: Drug: Sotatercept; Drug: vasodilator-based PAH therapy
- vasodilator-based PAH therapy alone (Active Comparator)
  Interventions: Drug: vasodilator-based PAH therapy

INTERVENTIONS:
Drug: Sotatercept — Sotatercept will be administered subcutaneously every 3 weeks for 24 weeks (total 8 injections): 0.3 mg/kg lead-in at Visit 1, then 0.7 mg/kg from Visit 2 if safety criteria are met. Dose holds/reductions follow label-concordant rules based on complete blood count (CBC) prior to each dose (e.g., hemoglobin rise >4.0 g/dL from baseline; or >2.0 g/dL from the previous dose and above ULN; or >2.0 g/dL above ULN; and platelet count <50,000/µL). Participants continue stable background PAH therapy (endothelin, nitric-oxide, prostacyclin pathways) per protocol; initiation or up-titration of PAH drugs during the 24-week treatment period is generally not permitted unless clinically mandated for safety and recorded as a protocol deviation.
  Arms: Sotatercept add-on + vasodilator-based PAH therapy
Drug: vasodilator-based PAH therapy — Participants receive no sotatercept. They continue site-standard, stable PAH therapy for 24 weeks (endothelin receptor antagonist, PDE5 inhibitor/riociguat, and/or prostacyclin class as clinically indicated). Changes to background therapy are discouraged during the 24-week period unless required for safety; any changes are captured for analysis. The same visit schedule and assessments (e.g., 6-minute walk test, biomarkers, clinical events) apply as in the sotatercept arm.

SUMMARY:
What is this study about? This study will test whether adding sotatercept to usual medicines for pulmonary arterial hypertension (PAH) can help adults who have PAH due to unrepaired congenital heart defects (atrial or ventricular septal defect, or patent ductus arteriosus), including Eisenmenger syndrome. These conditions often cause long-standing changes in the lung blood vessels and low oxygen levels.

Who can join? About 36 adults (age ≥18 years) in Japan whose PAH has not improved enough with pulmonary vasodilators may join. People with very severe symptoms (WHO class IV) or other serious illnesses will not be enrolled.

What will happen if I join?

Participants will be randomly assigned (like a coin flip, in a 2:1 ratio) to:

Sotatercept + vasodilator-based PAH care, or

vasodilator-based PAH care alone. The study lasts 24 weeks. Those who receive sotatercept will have injections every 3 weeks. All participants will have clinic visits and tests at the start, week 12, and week 24, including a 6-minute walk test (how far you can walk in 6 minutes), blood tests, questionnaires, and other heart-lung assessments used in routine PAH care.

What are the possible benefits? Sotatercept improved exercise capacity and heart-lung measures in other PAH studies, but people with unrepaired heart defects were not included. This study may or may not help you directly, but it may help doctors learn how to use sotatercept safely in this group.

What are the possible risks? Side effects seen with sotatercept include increase in haemoglobin, low platelets, nosebleeds, telangiectasia (small dilated blood vessels), bleeding, and blood clots. People with Eisenmenger syndrome can have both bleeding (for example, haemoptysis) and clotting risks. The study will check complete blood counts (CBC) regularly and adjust or pause dosing using label-based rules. Other risks are those of standard PAH care and blood tests.

Time and location The study is conducted at multiple hospitals in Japan. Study participation lasts about 6 months.

Costs and payments The study drug and study-specific tests will be provided at no cost. Usual medical care not required by the study will follow each hospital's standard billing. There is no required payment to join. Any travel reimbursement or stipends will follow site policy.

Privacy Your information will be kept confidential. Results will be shared in journals and at meetings without using your name.

Who to contact If you are interested or have questions, please contact the study team at the participating hospital.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years)
* unrepaired ASD, VSD or PDA
* ≥90 days of pulmonary vasodilator therapy; and either (i) pulmonary vascular resistance (PVR) ≥5 Wood units and mean pulmonary arterial pressure (mPAP) > 20 mm Hg on right heart catheterization within 180 days, or (ii) echocardiographic tricuspid regurgitation velocity >3.4 m/s with right-to-left/bidirectional shunt plus resting SpO₂ ≤92% consistent with cyanosis
* baseline 6MWD ≥100 m
* ability to complete questionnaires

Exclusion Criteria:

* WHO functional class IV; other unrepaired intracardiac shunts
* severe renal/hepatic/parenchymal lung disease or LVEF <40%
* prior sotatercept use
* contraindication to sotatercept per label
* investigator-judged unsuitability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance at 24 weeks from baseline | 24 weeks

SECONDARY OUTCOMES:
Mortality or lung transplantation | 24 weeks
PH-related hospitalisation or initiation of parenteral prostacyclin | 24 weeks
Change in WHO functional class at 24-week from baseline | 24 weeks
  A higher score indicates more severe symptom
Change in NT-pro BNP at 24-week from baseline | 24 weeks
Change in emPHasis-10 at 24-week from baseline | 24 weeks
  A higher score indicates more severe symptom

OTHER OUTCOMES:
PAH specific genetic test | 0 week
Changes in blood pressure (systolic and diastolic) | 0, 12, 24 weeks
  Office resting BP
Changes in pulse rate | 0, 12, 24 weeks
  bpm
Changes in oxygen saturation | 0, 12, 24 weeks
  Pulse Oxygen Saturation (Office, Resting)
Changes in hemoglobin | 0, 12, 24 weeks
  g per dL
Changes in platlet counts | 0, 12, 24 weeks
Changes in catheter-based mPAP | 0, 24 weeks
  mm Hg
Changes in catheter-based PVR | 0, 24 weeks
  Wood units
Changes in catheter-based Qp/Qs | 0, 24 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Kyushu University Hospital, Fukuoka, Not Required For This Country
  - The Second Department of Internal Medicine, University of Occupational and Environmental Health, Fukuoka
  - Division of Cardiovascular Medicine, Kobe University Hospital, Kobe
  - Department of Cardiovascular Medicine, Graduate School of Medical Science, Kyoto Prefectural University of Medicine, Kyoto
  - Department of Cardiology, Nagoya University Hospital, Nagoya
  - Department of Cardiovascular Medicine, Faculty of Medicine, Dentistry and Pharmaceutical Sciences, Okayama University, Okayama
  - Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine, Sendai
  - Department of Cardiology, Keio University School of Medicine, Tokyo
  - Department of Cardiovascular Medicine, Kyorin University School of Medicine, Tokyo
  - Division of Cardiovascular Medicine, Department of Internal Medicine, Showa University Graduate School of Medicine, Tokyo

IPD SHARING:
Plan to Share IPD: No